CLINICAL TRIAL: NCT05000866
Title: Expanding the Potential of Couples HIV Testing: Adjunct Modules to Reduce Drug Use Among Vulnerable Male Couples
Acronym: 4Us
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Tyrel Starks, Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA050508 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-08-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Substance Use; HIV Infections
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections

STUDY DESIGN:
Intervention Model Description: This study utilizes a randomized controlled trial design to evaluate the efficacy of two intervention components for couples HIV testing and counseling (CHTC): a communication skills training video and a substance use module. Participants are randomized in a full-factorial design to one of 4 conditions: CHTC as usual; CHTC + communication skills training videos; CHTC + substance use module; or CHTC plus both adjunct components.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CHTC as usual (No Intervention): Participants complete the standard Couples HIV Testing and Counseling session (CHTC).
- CHTC and communications skills training video (Active Comparator): Participants complete the standard Couples HIV Testing and Counseling session and also watch a communication skills training video together.
  Interventions: Behavioral: Communication skills training video
- CHTC and substance use module (Active Comparator): Participants complete the standard Couples HIV Testing and Counseling session and also complete a substance use module together.
  Interventions: Behavioral: Drug use module
- CHTC, communications skills training and substance use module (Active Comparator): Participants complete the standard Couples HIV Testing and Counseling session and watch a communication skills training video and complete a substance use module together.
  Interventions: Behavioral: Communication skills training video; Behavioral: Drug use module

INTERVENTIONS:
Behavioral: Communication skills training video — The communication skills training video component is designed to be self-delivered. Four couples are depicted in separate scenes discussing HIV testing, drug use, sexual agreements, and drug use during sex. Each scene is viewed twice. In the initial viewing, the couple in the video makes one or more communication errors. The scene is subsequently viewed a second time and the couple utilizes more effective communication skills, resulting in a more adaptive resolution. Each scene is introduced by a narrator who points out communication errors and orients viewers to skills utilized in adaptive versions of each scene.
  Arms: CHTC and communications skills training video; CHTC, communications skills training and substance use module
Behavioral: Drug use module — The substance use module is administered after step 5 of CHTC and prior to the delivery of rapid HIV-test results. The couple was first asked to fill in a calendar for the past 30 days, indicating each day on which either member used drugs or consumed alcohol. Completion of the calendar is done through an ACCESS database to facilitate remote intervention delivery. After completion of the calendar, the HIV tester asked a series of debriefing questions designed to elicit the couples' perspective on their use, establish the couple's goals and limits for drug use, and make plans to achieve these goals.
  Arms: CHTC and substance use module; CHTC, communications skills training and substance use module

SUMMARY:
This study utilizes a randomized controlled trial design to evaluate the efficacy of two intervention components for couples HIV testing and counseling (CHTC): a communication skills training video and a substance use module. Participants are randomized in a full-factorial design to one of 4 conditions: CHTC as usual; CHTC + communication skills training videos; CHTC + substance use module; or CHTC plus both adjunct components.

ELIGIBILITY:
Inclusion Criteria:

* · Have a main partner who is another male and have been in a relationship for 3 month or longer

  * One participant must be between 17 and 29; Main partner can be any age above 17.
  * One participant must be HIV negative (as confirmed by rapid test)
  * One participant must have used at least 1 drug in the past 90 days (cocaine/crack, opiates, misuse of prescription medication, stimulants, psychedelics, ecstasy, ketamine, GHB)
  * One participant must have engaged in Transmission Risk Behavior (TRB) in the past 90 days

    o Defined as Condom-less Anal Sex (CAS) with a casual partner and/or CAS with a non-monogamous or serodiscordant main partner
  * Live in the NYC or Detroit metropolitan area
  * Speak English

Exclusion Criteria:

* · Any signs of serious mental illness or cognitive deficit

  * History of IPV with their main partner and safety concerns in the current relationship.

Ages: 17 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Both partners in the couple must identify as male.
Enrollment: 484 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Drug use frequency | 12 months
  Number of reported days of illicit drug use (amphetamines, cocaine/crack, GHB, ketamine or ecstasy) reported on quarterly timeline follow-back assessments
Urine assay for drug use | 12 months
  Positive urine screen for drug use assessed bi-annually
CAS with casual partners | 12 months
  Number of total anal sex acts (insertive and receptive) with casual partners reported on quarterly timeline follow-back assessments
Bacterial STI's | 12 months
  Any chlamydia or gonorrhea diagnosis assessed bi-annually

SECONDARY OUTCOMES:
Binge drinking | 12 months
  Number of days on which 5 or more drinks containing alcohol were reported on the quarterly timeline follow-back interview
Syphilis infection | 12 months
  Reactive RPR test assessed bi-annually
PrEP Uptake | 12 months
  self-reported receipt of a PrEP-prescription
PrEP adherence | 12 months
  taking 4 or more doses weekly as prescribed reported on quarterly timeline follow-back assessments

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Hunter College, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Starks TJ, D Kyre K, B Cowles C, Castiblanco J, Washington C, N Parker J, M Kahle E, Stephenson R. A full-factorial randomized controlled trial of adjunct couples HIV testing and counseling components addressing drug use and communication skills among sexual minority male couples. BMC Public Health. 2021 Nov 24;21(1):2158. doi: 10.1186/s12889-021-12208-3. PMID 34819058